CLINICAL TRIAL: NCT04109872
Title: Lenalidomide Observational Study in Patients With Mantle Lymphoma in Relapse/Refraction. Spanish Programme RRMCL Results.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-LEN-2018-01
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Lenalidomide; Mantle Cell Lymphoma; Relapsed; Refractory; RRMCL spanish program
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mantle cell lymphoma treated with lenalidomide cohort: Patients diagnosed with mantle cell lymphoma treated with leanalidomide through the RRMCL spanish program.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide effectiveness and tolerability data analysis, that will be retrospectively collected until the 30 of April 2018.

SUMMARY:
This is a multicentric, observational and retrospective study of the use of lenalidomide in patients with relapsed or refractory mantle cell lymphoma that are included in the RRMCL spanish program.

The lenalidomide effectiveness and tolerability data will be retrospectely collected until the 30 of April 2018.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Diagnosed with relapsed or refractory mantle cell lymphoma verified by a tissue biopsy.
* Treated with monotherapy or combination of lenalidomide.
* Not candidate for any of the therapeutic options approved until that date for this disease.
* Not candidate or unable to be included in any clinical trial due to availability or geographical difficulty.
* Registered in the RRMCL spanish program.

Exclusion Criteria:

* ECOG > 2.
* Patients with uncontrolled comorbidities.
* Blastoid variant.
* Central nervous system tumor infiltration.
* HIV, HBV and/or HCV active infection.
* Radiotherapy concomitant treatment or that have received radiotherapy in the previous 30 days to the beginning of the first cycle of lenalidomide.
* Diagnosed with other active solid tumor except for basal cell carcinoma skin cancer.
* Patients that haven´t completed at least one complete cycle of the treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with mantle cell lymphoma that received lenalidomide through the RRMCL program as long as they meet all the inclusion criteria and none of the exclusion and independently from being dead or alive in the moment of data record.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Experience of real clinal practice lenalidomide use. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  Results of the the usage in real clinical practice of the lenalidomide monotherapy or combination treatment in patients with relapsed or refractory mantle cell lymphoma that aren´t candidate to other alternative treatments inside the RRMCL spanish program.

SECONDARY OUTCOMES:
Proportion of patients that achieve objective response. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  The objective response will be measured in terms of complete response, not confirmed complete response and partial response according to the 2007 International Working Group criteria after the 6º treatment cycle.
Duration of the response. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  Partial and complete response duration.
Verify the disease free survival. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  The disease free survival is defined as the time that passes from the inclusion in the record until a control is done or takes place a relapse (local or distant).
Verify the disease overall survival. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  The disease overall survival is defined as the time that passes from the inclusion in the record until a control is done or the patient´s death.
Evaluate the incidence of treatment adverse events. | Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2019), whichever occurred first
  Number and description of adverse effects due to the lenalidomide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos García Pérez, Study Chair — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain